CLINICAL TRIAL: NCT04823494
Title: Protocol for Self-Fitting Hearing Aid Wear-Time Trial for Listeners With Mild to Moderate Hearing Loss
Brief Title: Wear-Time Trial for Self-Fitting Hearing Aid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GN Hearing A/S (Industry)
Collaborators: Northwestern University (Other); Sertoma Speech and Hearing Center (Other); Vanderbilt University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: X-Men
Record Dates: First submitted 2021-03-26; First posted 2021-03-30 (Actual); Results first posted 2022-05-11 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-03

CONDITIONS: Hearing Loss, Sensorineural
MeSH Terms: conditions — Hearing Loss, Sensorineural | interventions — Hearing Aids

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Pro-Fit followed by Self Fit (Experimental): Hearing aids fit by a professional hearing care provider using best practices followed by patient ...
  Interventions: Device: Hearing aids
- Self-Fit followed by ProFit (Experimental): Hearing aids fit by patient followed by ...
  Interventions: Device: Hearing aids

INTERVENTIONS:
Device: Hearing aids — Earbud style hearing aids fit to both ears

SUMMARY:
This document describes a clinical validation study for a double-blind repeated-measures comparative study of the Great Nordic (GN) self-fitting method to a validated audiology-best-practices method when fitting the GN Self-fitting Hearing Aid, a device intended for persons aged 18-75 years old who have mild-to-moderate hearing loss. A crossover wear-time field trial will be conducted. The focus of the study is on the validity of the self-fitting process used to select appropriate frequency-gain characteristics for the GN Self-fitting Hearing Aid, and the safety and effectiveness of the device.

ELIGIBILITY:
Inclusion Criteria:

* Mild-to-moderate bilateral sensorineural hearing loss (thresholds from 250 - 8000 Hz less than 60 decibels Hearing Level (dB HL) and from 2000 - 8000 Hz, at least one threshold greater than 20 dB HL)
* Mix of male and female subjects (aiming for a representative balance)
* Mix of prior hearing-aid use (aiming for 70-80% persons with no prior hearing aid use)
* 18-75 years old (aiming for primarily 50-70 years old, with avg. age ~65 years)
* Apple iPhone (iOS 14 compatible or greater, as required for the SELF-FIT app)
* Able to read and comprehend English
* Patient willing to provide informed consent

Exclusion Criteria:

* Hearing outside of limits noted above
* Self-reported ear-related pathology (including chronic severe dizziness or chronic severe tinnitus)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-06-18 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd Ricketts, Ph.D., Principal Investigator — Vanderbilt University; Sumitrajit Dhar, Ph.D., Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Sertoma Speech and Hearing Center, Palos Hills, Illinois
  - Vanderbilt University, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cox RM, Alexander GC. The abbreviated profile of hearing aid benefit. Ear Hear. 1995 Apr;16(2):176-86. doi: 10.1097/00003446-199504000-00005. PMID 7789669
- [Background] Killion MC, Niquette PA, Gudmundsen GI, Revit LJ, Banerjee S. Development of a quick speech-in-noise test for measuring signal-to-noise ratio loss in normal-hearing and hearing-impaired listeners. J Acoust Soc Am. 2004 Oct;116(4 Pt 1):2395-405. doi: 10.1121/1.1784440. PMID 15532670

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Visit 1 included tests to determine study eligibility and baseline (unaided) performance for outcomes measures obtained after each segment of the crossover field trial (Visits 2 and 3). Eligible subjects were assigned successively to one of two treatment orders at each site for counterbalancing of treatment order. As a result, all 40 enrollees met selection criteria and were assigned to one of the two treatment orders.
Groups:
- Pro-Fit Followed by Self-Fit: Hearing aids fit by a professional hearing care provider using best practices, followed by a self-fit of both devices. There was a 10-14-day wear period following each fitting method.
  Hearing aids: Earbud style hearing aids fit to both ears
- Self-Fit Followed by Pro-Fit: Hearing aids self-fit by participant followed by the fitting of the devices by a professional hearing care provider using best practices. There was a 10-14-day wear period following each fitting method.
  Hearing aids: Earbud style hearing aids fit to both ears
Period: Overall Study
Arm/Group | Pro-Fit Followed by Self-Fit | Self-Fit Followed by Pro-Fit
Started | 21 | 19
Completed | 19 | 18
Not Completed | 2 | 1
Not completed — Programming software malfunction. | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Devices lost | 0 | 1

BASELINE CHARACTERISTICS:
Population: 37 subjects completed both Pro-Fit and Self-Fit conditions in a counterbalanced order. Subjects switched conditions after the first of two wear time trials. There were a total of 37 subjects tested.
Groups:
- Pro-Fit Followed by Self-Fit: Hearing aids initially fit by a professional hearing care provider using best practices and worn for 10-14 days. Devices then self-fit by participant and worn for 10-14 days.
  Hearing aids: Earbud style hearing aids fit to both ears
- Self-Fit Followed by Pro-Fit: Hearing aids self-fit by patient initially and worn for 10-14 days. Devices then fit by a professional hearing care provider using best practices and worn for another 10-14 days.
  Hearing aids: Earbud style hearing aids fit to both ears
- Total: Total of all reporting groups
Arm/Group | Pro-Fit Followed by Self-Fit | Self-Fit Followed by Pro-Fit | Total
Number analyzed (Participants) | 19 | 18 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 8 | 19
  >=65 years | 8 | 10 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.95 (8.71) | 58.67 (15.11) | 59.84 (12.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 10 | 9 | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 18 | 37

OUTCOME MEASURES:

1. Primary Outcome: Aided Abbreviated Profile of Hearing Aid Benefit (APHAB)
Description: The APHAB is a 24-item self-assessment of the amount of trouble the respondent has with communication in everyday situations. Sample question: "When I'm at the dinner table with several people, and I am trying to have a conversation with one person, understanding speech is difficult." For each of the 24 items, person asked to select one of the following percentages to indicate how frequently this occurs: Always (99%); Almost Always (87%); Generally (75%); Half-the-time (50%); Occasionally (25%); Seldom (12%); or Never (1%). Mean scale scores are expressed as a percentage or proportion representing the average frequency of difficulty experienced. An APHAB global score based on the 18 items from the three speech-communication subscales was used in the statistical analyses. APHAB scores were obtained unaided (Visit 1) and following use of the hearing aids for 10-14 days for each fit (Visits 2 & 3; aided). The primary outcome is the mean difference in aided scores, Self-Fit minus Pro-Fit.
Time Frame: 10-14 days
Population: Crossover design. All 37 subjects participated in both Pro-Fit and Self-Fit phases with about half receiving each intervention first. Subjects crossed after 10-14 day field use.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Pro-Fit: Hearing aids fit by a professional hearing care provider using best practices and worn for 10-14 days prior to outcomes measurement.
  Hearing aids: Earbud style hearing aids fit to both ears
- Self-Fit: Hearing aids self-fit by participant and worn 10-14 days prior to outcomes measurement.
  Hearing aids: Earbud style hearing aids fit to both ears
Arm/Group | Pro-Fit | Self-Fit
Number analyzed (Participants) | 37 | 37
score on a scale | 21.35 [16.78 to 26.33] | 22.76 [18.33 to 27.59]
Statistical Analysis 1: Comparison: Pro-Fit vs Self-Fit; For the wear-time crossover field trial, the APHAB was measured following both the audiology best-practices hearing aid fitting (PRO-FIT) and the self-fitting method (SELF-FIT). * Null hypothesis: Mean (APHAB SELF-FIT - APHAB PRO-FIT ) ≥ 8.4 * Alternative hypothesis: Mean (APHAB SELF-FIT - APHAB PRO-FIT) < 8.4 The mean difference between the aided scores for the two fitting methods, Self-Fit minus Pro-Fit, represent the primary outcome measure. The expected difference = 0; Test type: Non-Inferiority — For sample size in each sequence group is 16 (total N=32), a 2 X 2 crossover design will have 80% power to reject the null hypothesis that the SELF-FIT APHAB mean is inferior to the PRO-FIT APHAB mean. The non-inferiority difference margin is 8.4, the standard deviation of differences is 16.3, and p<.025. The non-inferiority margin of 8.4 preserves half the 95% critical difference for the global APHAB score (16.8). The common standard deviation reported for the APHAB global score is 16.0; p < 0.025, t-test, 1 sided — There were two outcome measures, primary and secondary, considered. As a result, the a priori p value of .05 for statistical significance was adjusted for multiple comparisons to .025; The mean differences and 95% CIs in APHAB global score between SELF-FIT and PRO-FIT were calculated using bias-corrected & accelerated bootstrapping; Mean Difference (Final Values) = 1.4, 95% CI 2-sided [-1.59 to 4.73] — The mean difference and 95% CIs are for Self-Fit minus Pro-Fit aided scores. These values are the pooled data for all 37 participants, 19 receiving one sequence and 18 the other sequence

2. Secondary Outcome: Quick Speech in Noise Test (QuickSIN)
Description: The QuickSIN test consists of lists of six sentences played from a loudspeaker at a constant level approximating typical conversation. The level of the co-located four-talker babble (background noise) increased across the six sentences for signal-to-noise ratios (SNRs) ranging from +25 to 0 decibels (dB) SNR (in steps of 5 dB). The participant was asked to repeat each sentence. The examiner scored predetermined key words in each sentence. The resulting score was interpreted as an SNR loss in dB where a value near 0 dB indicates normal hearing and larger values indicate more difficulty listening in noise. The QuickSIN SNR values for the Pro-Fit condition were subtracted from those for the Self-Fit condition to generate a difference value in dB between the two fitting methods. The secondary outcome measure evaluated here was the mean difference in QuickSIN SNR values in dB between Pro-Fit and Self-Fit for all 37 participants; 19 Pro-Fit first and 18 Self-Fit first.
Time Frame: Measurement after 10-14-day wear time for each fit.
Population: Crossover design. All 37 subjects participated in both Pro-Fit and Self-Fit phases. Subjects crossed after 10-14 day field use.
Measure: Mean (95% Confidence Interval); unit: score on a scale (dB)
Groups:
- Pro-Fit: Hearing aids fit by a professional hearing care provider using best practices and worn for 10-14 days.
  Hearing aids: Earbud style hearing aids fit to both ears
- Self-Fit: Hearing aids fit by participants and worn for 10-14 days.
  Hearing aids: Earbud style hearing aids fit to both ears
Arm/Group | Pro-Fit | Self-Fit
Number analyzed (Participants) | 37 | 37
score on a scale (dB) | 2.19 [1.53 to 2.89] | 2.77 [2.18 to 3.37]
Statistical Analysis 1: Comparison: Pro-Fit vs Self-Fit; For the QuickSIN, aided performance after each wear period was compared between SELF-FIT and PRO-FIT. * Null hypothesis: Mean (QuickSIN SELF-FIT - QuickSIPRO-FIT) ≥ 1.5 dB * Alternative hypothesis: Mean (QuickSIN SELF-FIT - QuickSIN PRO-FIT) < 1.5 dB Power calculations were based on the primary outcome measured, the aided APHAB global score, (see information for that outcome measure). With the minimum required N of 32 based on the APHAB global score, the power for QuickSIN exceeded 80%; Test type: Non-Inferiority — For the QuickSIN, a clinically meaningful difference is 3 dB and half that difference resulted in a margin of 1.5 dB. This 1.5-dB margin was used for the QuickSIN for the non-inferiority analyses of the data from the field-trial component. The mean difference, QuickSIN Self-Fit minus QuickSIN Pro-Fit, should be less than 1.5 dB for the entire sample (N=37) to meet the non-inferiority criterion; p < 0.025, t-test, 1 sided — The a priori threshold value of 0.05 was Bonferroni-adjusted to 0.025 based on the use of two outcome measures, APHAB global (primary) and QuickSIN (secondary); The mean differences in dB, SELF-FIT minus PRO-FIT, were calculated with 95% confidence intervals (bias-corrected, accelerated bootstrap) generated; Mean Difference (Final Values) = 0.58, 95% CI 2-sided [-0.03 to 1.20] — Mean differences in aided QuickSIN SNR in dB, Self-Fit minus Pro-Fit, were calculated for the entire group of 37 participants with about 1/2 receiving one of the two fit sequences (Pro-Fit then Self-Fit or Self-Fit then Pro-Fit)

ADVERSE EVENTS:
Time Frame: The time from eligibility and baseline measures at Visit 1 through the completion of the outcome measures after the second wear period was 3-5 weeks. Adverse events were collected over this time frame for each participant.
Description: One potential adverse effect was an adjustment of gain that could result in uncomfortable loudness. However, this was prevented automatically for all participants by limiting the maximum output of the devices.
  The app used to fit and control the device requires some familiarity with apps and the user may experience some frustration with these procedures initially.
  Adverse events and serious adverse events were monitored throughout the study for all participants. None were recorded.
Groups:
- Self-Fit: Hearing aids self-fit by participant and worn for 10-14 days.
  Hearing aids: Earbud style hearing aids fit to both ears
Arm/Group | Pro-Fit | Self-Fit
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/37
Other Adverse Events (participants affected / at risk) | 0/37 | 0/37

LIMITATIONS AND CAVEATS:
The minimum N needed to achieve the desired statistical power was 32 and 40 participants were enrolled to allow for attrition. In the end, only 3 participants were exited from the study or withdrew, leaving 37 with complete data. Of the 3 with incomplete data, 2 resulted from technical issues with the devices or app. However, both per-protocol analyses (summarized above) and intention-to-treat analyses yielded the same findings, indicating that the few missing data were inconsequential.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-03): https://cdn.clinicaltrials.gov/large-docs/94/NCT04823494/Prot_SAP_000.pdf